CLINICAL TRIAL: NCT03096249
Title: Monitoring the Influence of Oxytocin on Socio-communicative Sensitivity Using Fast Periodic Visual Stimulation
Brief Title: The Influence of Oxytocin on Socio-communicative Sensitivity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SingleOT_EEG_S56327
Record Dates: First submitted 2017-03-07; First posted 2017-03-30 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Oxytocin
Keywords: oxytocin; emotion recognition; emotion processing; social salience; face processing; Electroencephalography (EEG)
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Syntocinon nasal spray (40 IU/ml; oxytocin, product code RVG 03716) will be used for intranasal administration of a single intranasal dose of 24 international units (IU; 3 puffs of 4 IU per nostril)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Physiological water (sodium chloride (NaCl) solution) Administration via nasal spray
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — Syntocinon nasal spray: single dose of 24IU (3 puffs of 4IU per nostril)
  Arms: Oxytocin
Other: Placebo — Placebo spray: single dose (3 puffs per nostril).
  Arms: Placebo

SUMMARY:
Oxytocin (OT) is a neuropeptide that acts as a neurotransmitter and neuromodulator in the brain. Previous studies have shown that intranasal administration of OT improves social cognition and behavior (e.g. emotion recognition). In the current study, we want to gain more insight into the underlying mechanisms by which OT influences emotion recognition. More specifically, we will investigate whether intranasal administration of OT enhances the salience of social (compared to non-social) information and whether it increases the neural sensitivity for subtle socio-emotional cues, by recording scalp electroencephalography (EEG) during Fast Periodic Visual Stimulation (FPVS).

DETAILED DESCRIPTION:
The present study is a double-blind, randomized, placebo-controlled, crossover clinical trial, in which (approximately 30) neurotypical male adults (18 to 30 years old) will participate. All participants will perform two sessions (OT and placebo), separated by two weeks. For the first session, the participants are randomly assigned to the placebo or the OT condition. Syntocinon nasal spray will be used for intranasal administration.

In each session, we will measure the neural salience/sensitivity for socio-emotional information, by recording EEG during FPVS. Participants simply have to press a button when the fixation cross turns red, while watching rapidly alternating visual stimuli. Starting 20 minutes after substance intake, four FPVS paradigms are administered in randomized order:

1. A frequency-tagging FPVS paradigm, to measure the salience of social versus non-social stimuli.
2. The oddball face detection paradigm, to assess the neural sensitivity to faces embedded in a series of objects.
3. The oddball identity discrimination task, to examine the ability to discriminate between faces with a different identity.
4. The oddball expression generalization task, to investigate the sensitivity for facial emotional expressions embedded within neutral faces with varying identities.

After two FPVS paradigms, a four minutes resting state EEG measure will be performed. At the end of the session, emotion recognition will be measures with the Palermo matching task (65 items).

The primary aim is to investigate whether the performance on each of these paradigms/tasks differs between the OT and the placebo condition. Furthermore, we want to explore whether the effect of OT is influenced by the participant's attachment style, social responsiveness, social phobia, or mood, which will be assessed via self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 30 years
* male
* right-handed
* typically developing
* Normal or adjusted-to-normal vision (with glasses or lenses)

Exclusion Criteria:

* psychiatric disorder
* neurological disorder (e.g. epilepsy, migraine)
* color blindness
* psychoactive medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
social salience frequency-tagging FPVS | random: 30-70 minutes after nasal spray
  EEG recording during simultaneous (superimposed) presentation of social stimuli (faces) and non-social stimuli (objects or houses), at a frequency of 6 and 7.5Hz, respectively (counterbalanced).
Oddball face detection FPVS paradigm | random: 30-70 minutes after nasal spray
  EEG recording during presentation of objects (at 6 Hz) and faces (inserted as an "oddball" every fifth image, thus at a frequency of 1.2 Hz)
Oddball identity discrimination FPVS paradigm | random: 30-70 minutes after nasal spray
  EEG recording during presentation of neutral faces of the same person (same identity, presented at 6 Hz) and the face of another person (inserted as an "oddball" every fifth image, thus at a frequency of 1.2 Hz)
Oddball expression generalization FPVS paradigm | random: 30-70 minutes after nasal spray
  EEG recording during presentation of neutral faces with different identities (at 6 Hz) and faces with an emotional expression (fear, anger, happy; inserted as an "oddball" every fifth image, thus at a frequency of 1.2 Hz)

SECONDARY OUTCOMES:
Emotion recognition: accuracy on the Palermo Matching task (65 items) | 80 minutes after nasal spray (after all EEG measures)
  Three faces are shown on the screen. Two of them display the same emotion and the participant has to indicate which face shows a different emotion
resting state EEG | 45-50 minutes after nasal spray (after two FPVS paradigms)
  EEG recording, while presenting a fixation cross
Social responsiveness: Social Responsiveness Scale (SRS) | Baseline
  Self-report version of the SRS. In addition to a Total score reflecting severity of social deficits in the autism spectrum, the SRS generates scores for five Treatment subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behavior.
Social phobia: Social Phobia Inventory (SPIN) | Baseline
  A 17-item questionnaire that screens for, and measures, the severity of social anxiety disorder.
Attachment: State Adult Attachment Measure (SAAM) | Baseline
  The SAAM measures 3 different aspects of adult attachment: Security, Anxiety, Avoidance. There are 21 Likert-style questions with a score between 1 and 7 (7 for each of the three subscales).
Mood: Positive And Negative Affect Schedule (PANAS) | 90 minutes after nasal spray
  The Positive and Negative Affect Schedule (PANAS) comprises two mood scales, one that measures positive affect and the other which measures negative affect. It consists of 20 items (10 for each subscale).

OTHER OUTCOMES:
side-effect questionnaire | 90 minutes after nasal spray

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, Professor, Principal Investigator — KU Leuven (Catholic University Leuven)
Locations (1):
- Biomedical Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided